CLINICAL TRIAL: NCT06858696
Title: An Open-label, Non-randomized Study to Evaluate the Pharmacokinetics (PK), Safety and Tolerability of a Single Dose of Mavorixafor in Participants With Hepatic Impairment (HI) Compared to Matched Healthy Volunteers With Normal Hepatic Function
Brief Title: A Study to Investigate Pharmacokinetics (PK) and Safety of a Single Dose of Mavorixafor in Participants With Hepatic Impairment (HI) Compared to Matched Healthy Volunteers With Normal Hepatic Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-003
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — mavorixafor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: Child-Pugh A (Experimental): Participants with mild HI will receive a single dose of mavorixafor orally on an empty stomach, following a minimum 10-hour fasting period.
  Interventions: Drug: Mavorixafor
- Group 2: Child-Pugh B (Experimental): Participants with moderate HI will receive a single dose of mavorixafor orally on an empty stomach, following a minimum 10-hour fasting period.
  Interventions: Drug: Mavorixafor
- Group 3: Child-Pugh C (Experimental): Participants with severe HI will receive a single dose of mavorixafor orally on an empty stomach, following a minimum 10-hour fasting period.
  Interventions: Drug: Mavorixafor
- Group 4: HVs (Experimental): HVs matched with the mild HI participants will receive a single dose of mavorixafor orally on an empty stomach, following a minimum 10-hour fasting period.
  Interventions: Drug: Mavorixafor
- Group 5: HVs (Experimental): HVs matched with the moderate HI participants will receive a single dose of mavorixafor orally on an empty stomach, following a minimum 10-hour fasting period.
  Interventions: Drug: Mavorixafor
- Group 6: HVs (Experimental): HVs matched with the severe HI participants will receive a single dose of mavorixafor orally on an empty stomach, following a minimum 10-hour fasting period.
  Interventions: Drug: Mavorixafor

INTERVENTIONS:
Drug: Mavorixafor — Mavorixafor will be administered per schedule specified in the arm description.

SUMMARY:
The purpose of this study is to measure the effect of HI on the PK, safety, and tolerability of a single dose of mavorixafor compared to matched healthy volunteers (HVs) with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight is more than 50.0 kilograms (kg) with body mass index (BMI) between 18.0 and 40.0 kg/square meter (m^2) at the Screening Visit and at Day -1 Visit.
* In good health, as determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations.
* Current non-smoker or light smoker, that is, no more than 10 cigarettes or 10 milligrams (mg) equivalent use of nicotine per day by e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch, nicotine gum, and able and willing to refrain from smoking and tobacco use during the study.

Inclusion criteria applicable to participants with HI Only:

* Aside from hepatic insufficiency, the participant is deemed by the Investigator to be sufficiently healthy for study participation, based upon medical history, physical examination, vital signs, and screening laboratory evaluations.
* Documented chronic stable liver disease according to CP classification with diagnosis of HI due to parenchymal liver disease.
* Currently on a stable medication regimen, defined as not starting new drug(s) or changing drug dose(s) within 28 days of the mavorixafor administration (Day 1).

Key Exclusion Criteria:

* Female participants/volunteers who are breastfeeding or female participants/ volunteers with a positive pregnancy test at the Screening Visit or at Day -1.
* History of allergy to mavorixafor excipients or drugs in a similar pharmacological class with mavorixafor.
* Has an active malignancy or history (≤ 5 years prior to enrollment) of solid, metastatic, or hematologic malignancy.
* A known history of positive serology or viral load for human immunodeficiency virus (HIV) or a known history of acquired immunodeficiency syndrome.
* Known active COVID-19 infection or a positive test within the local accepted clinical and governmental guidelines for a communicable window.
* Positive hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb).
* Positive hepatitis C antibody test result at screening.
* Have received mavorixafor previously.
* Has used an investigational drug within 30 days (or 5 half-lives whichever is longer) before the first dose of mavorixafor.

Additional exclusion criteria applicable to Volunteers with Normal Hepatic Function Only:

* History or evidence of liver disease such as alcoholic liver disease, autoimmune hepatitis, hepatitis B, hepatitis C, primary biliary cirrhosis, primary sclerotic cholangitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug induced liver injury, and/or hepatocellular carcinoma.
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal, neurological, or psychiatric disorder.
* Clinical laboratory test results must be strictly within the normal laboratory reference ranges for liver function and hematology, and for other parameters, deemed as not clinically significant by the Investigator.

Additional exclusion criteria applicable to participants with HI Only:

* Clinically significant abnormal laboratory values at screening or Day -1, in the judgment of the Investigator.
* History of liver transplant or currently in the top 5% of recipients on the transplant list.
* Evidence of hepatorenal syndrome or abnormal serum creatinine levels (above upper limit for the local lab) and estimated glomerular filtration rate < 60 milliliters (mL)/minute (min) or abnormal sodium and potassium levels.
* New medication or a change in dose for hepatic encephalopathy within the 3 months prior to admission to the clinical site, unless approved by the Investigator and the study Medical Monitor.
* Concurrent conditions that could interfere with safety and/or tolerability measurements.

NOTE: Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Mavorixafor | Predose up to 192 hours postdose (Day 1 up to Day 9)
Area Under the Serum Concentration Curve From Time Zero to the Last Measurable Concentration (AUC0-last) of Mavorixafor | Predose up to 192 hours postdose (Day 1 up to Day 9)

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Day 15
Time to Reach Cmax (Tmax) of Mavorixafor | Predose up to 192 hours postdose (Day 1 up to Day 9)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — X4 Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Catalina Research Institute, LLC, Montclair, California
  - Catalina Research Institute, LLC, Rialto, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute/Alamo Medical Research, San Antonio, Texas